CLINICAL TRIAL: NCT03737071
Title: The Effects of Low Carbohydrate Diet on Liver Fat Content and Mitochondrial Fluxes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Panu Luukkonen, MD, PhD, Helsinki University Central Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HUS21372018
Record Dates: First submitted 2018-11-06; First posted 2018-11-09 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Fatty Liver
MeSH Terms: conditions — Fatty Liver | interventions — Diet, Carbohydrate-Restricted

STUDY DESIGN:
Intervention Model Description: Low Carbohydrate Diet versus Simple Calorie Restriction Diet
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Carbohydrate Diet (Experimental): Low Carbohydrate Diet
  Interventions: Behavioral: Low Carbohydrate Diet
- Simple Calorie Restriction Diet (Active Comparator): Simple Calorie Restriction Diet
  Interventions: Behavioral: Simple Calorie Restriction Diet

INTERVENTIONS:
Behavioral: Low Carbohydrate Diet — Ketogenic dietary intervention
  Arms: Low Carbohydrate Diet
Behavioral: Simple Calorie Restriction Diet — Simple calorie restriction dietary intervention
  Arms: Simple Calorie Restriction Diet

SUMMARY:
The purpose of this study is to examine whether a low carbohydrate diet as compared to simple calorie restriction decreases hepatic lipid content and changes hepatic mitochondrial flux in humans.

DETAILED DESCRIPTION:
In this study, the investigators will examine whether a low carbohydrate diet as compared to simple calorie restriction will change hepatic lipid content and mitochondrial flux in humans. Before and after a low carbohydrate diet and a simple calorie restriction intervention, rates of hepatic mitochondrial flux will be assessed using positional isotopomer analysis of 3-13C-lactate during a 3 hour basal period. Rates of whole body ketogenesis will be determined using [13C4]β-hydroxybutyrate, and whole body glucose metabolism will be measured using [2H7]glucose. Body composition will be determined with bioelectrical impedance; hepatic lipid content will be measured with MRS. Whole-body oxidation of lipids, carbohydrates and protein will be determined using indirect calorimetry.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70
* Subjects must be able to communicate meaningfully with the investigator and must be legally competent to provide written informed consent

Exclusion Criteria:

* chronic liver disease other than NAFLD
* chronic disease associated with hepatic steatosis such as diabetes mellitus
* use of drugs known to affect hepatic steatosis
* contraindications for MRI
* pregnancy or nursing at the time of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-11-15 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Change in hepatic triglyceride content | 1 week
  Change in hepatic triglyceride content will be measured using 1H magnetic resonance spectroscopy (MRS).
Change in hepatic mitochondrial flux | 1 week
  Change in the rate of hepatic mitochondrial flux (Vcs) will be assessed using 3-13C-lactate infusion.

SECONDARY OUTCOMES:
Change in beta-hydroxybutyrate production rate | 1 week
  Change in the rate of beta-hydroxybutyrate production will be assessed using [13C4]β-hydroxybutyrate infusion.
Change in glucose production rate | 1 week
  Change in the rate of glucose production will be assessed using [2H7]glucose infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Panu Luukkonen, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Biomedicum 2U, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: No
IPD will be shared as much as our ethics permission and the GDPR regulations of the European Union allow

REFERENCES:
- [Derived] Qadri SF, Porthan K, Dufour S, Lehtimaki TE, Petersen KF, Shulman GI, Yki-Jarvinen H, Luukkonen PK. Distinct effects of ketogenic and non-ketogenic weight-loss diets on hepatic steatosis and mitochondrial metabolism in MASLD. J Hepatol. 2026 Feb 6:S0168-8278(26)00062-0. doi: 10.1016/j.jhep.2026.02.001. Online ahead of print. PMID 41655910